CLINICAL TRIAL: NCT04072653
Title: Sentinel Node Biopsy Vs Observation After Axillary PET Examination
Brief Title: Sentinel Node Biopsy Vs Observation After Axillary PET
Acronym: SOAPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-SOAPET
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: In the first stage, the negative predictive value is evaluated in patients with negative preoperative axillary assessment, including LymphPET and routine imaging examinations. In the second stage, sentinel lymph node biopsy will be spared in the patients with negative preoperative axillary assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation group( SLNB is spared) (Experimental): In the second stage, sentinel lymph node biopsy will be spared in the patients with negative preoperative axillary assessment.
  Interventions: Procedure: SLNB is spared

INTERVENTIONS:
Procedure: SLNB is spared — SLNB is spared in patients with negative preoperative axillary assessment(including LymphPET and other imaging examinations)

SUMMARY:
Several researches have proved that avoiding axillary surgery does not worsen the outcome of breast cancer patients with relatively low risk. Based on the routine axillary imaging evaluation (ultrasound and MR etc.) and latest dedicate lymph node PET (LymphPET), axillary nodal burden can be identified before operation.

Therefore this prospective study are designed to evaluate the negative predictive value of LymphPET and to verify whether sentinel lymph node biopsy can be spared in patients with negative preoperative axillary assessment.

ELIGIBILITY:
Inclusion Criteria:

stage 1:

1. female
2. ≥18 years old
3. invasive ductal carcinoma or DCIS proved by core needle biopsy
4. tumor size ≤ 5cm
5. negative preoperative axillary assessment(including body examination, ultrasound and MR examination)
6. patients is accessible for the following axillary surgery and pathological test(including sentinel lymph node biopsy and axillary lymph node dissection)

stage 2:

1. female
2. ≥18 years old
3. invasive carcinoma proved by core needle biopsy
4. has plan for breast conserving surgery and adjuvant radiation after surgery
5. negative preoperative axillary assessment(including body examination, ultrasound and axillary PET mSUV<0.27)
6. patients is accessible for the follow up

Exclusion Criteria:

stage 1:

1. distant metastases
2. in the procedure of neoadjuvant therapy
3. positive preoperative axillary assessment (including body examination, ultrasound and MR examination)
4. pregnancy or breastfeeding
5. axillary biopsy or axillary surgery before LymphPET
6. suffer from diabetes mellitus and without well control of bloodglucose
7. previous malignancy
8. allergic to tracer of LymphPET

stage 2:

1. distant metastases
2. in the procedure of neoadjuvant therapy
3. positive preoperative axillary assessment (including body examination, ultrasound and PET mSUV≥0.27)
4. pregnancy or breastfeeding
5. axillary biopsy or axillary surgery before LymphPET
6. suffer from diabetes mellitus and without well control of bloodglucose
7. previous malignancy
8. allergic to tracer of LymphPET

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1528 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
stage 1: negative predictive value | 6 months
  negative predictive value of LymphPET in breast cancer patients with a negative preoperative axillary assessment
stage 2: D-DFS(distant disease-free survival) | 5 years
  D-DFS of patients with negative preoperative axillary assessment(including LymphPET and other imaging examination) and for whom axillary surgery is spared
stage 2: LRFS(local-regional free survival) | 5 years
  LRFS of patients with negative preoperative axillary assessment(including LymphPET and other imaging examination) and for whom axillary surgery is spared

SECONDARY OUTCOMES:
stage 1: false negative rate | 6 months
  false negative rate of LymphPET in breast cancer patients with a negative preoperative axillary assessment
stage 2: DFS(disease-free survival) | 5 years
  DFS of patients with negative preoperative axillary assessment(including LymphPET and other imaging examination) and for whom axillary surgery is spared
stage 2: OS(overall survival) | 5 years
  OS of patients with negative preoperative axillary assessment(including LymphPET and other imaging examination) and for whom axillary surgery is spared
stage 2: adverse events of upper limbs | 5 years
  adverse events of patients with negative preoperative axillary assessment(including LymphPET and other imaging examination) and for whom axillary surgery is spared，as assessed by CTCAE v5.0
stage 2: breast self evaluation | 5 years
  breast self evaluation for patients with negative preoperative axillary and for whom axillary surgery is spared, as assessed by BREAST Q© index. The BREAST-Q has a modular, procedure-specific structure with scales that evaluate both satisfaction and quality of life. Psychometric evaluation reveals high reliability, validity and responsiveness to surgical intervention across all scales. Breast Q is composed of aesthetical and emotional modules, and each score ranges from 1 to 4 points (higher values represent a better self evaluation). By comparing the sum of the score in different modules before and after the surgery, Breast Q can help to facilitate a self evaluation for breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Min Shao, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No